CLINICAL TRIAL: NCT01423682
Title: The Influence of Eccentric Training on the Volume and Vascularisation of the Rotator Cuff in Patients With Rotator Cuff Tendinopathy and Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: Fund for Scientific Research, Flanders, Belgium (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2011/482
Record Dates: First submitted 2011-08-23; First posted 2011-08-26 (Estimated); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Rotator Cuff Tendinopathy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy subjects (Placebo Comparator)
  Interventions: Behavioral: Eccentric exercise
- Rotator cuff tendinopathy (Active Comparator)
  Interventions: Behavioral: Eccentric exercise

INTERVENTIONS:
Behavioral: Eccentric exercise — Patients and healthy subjects will perform an eccentric exercise during which a weight is lifted along the body and lowered with an extended arm at a slow speed. Weight is determined, based on pain in patients and based on force in healthy subjects.

SUMMARY:
Patients with rotator cuff tendinopathy make up a large part of the population in physiotherapy practice. The rotator cuff, a shoulder muscle group, plays an important role in causing pain. Tendons suffer large compression and friction, which can lead to degeneration of these tendons. Rehabilitation often leads to unsatisfying results.

In Achilles and patella tendinopathy, a new training program called eccentric training has shown very good results. Eccentric training contains exercises during which a force has to be resisted while the muscle lengthens instead of shortens. This would have a larger influence on tendon tissue. Some small studies also show promising results of eccentric training in patients with rotator cuff tendinopathy but the mechanisms behind these results remain unclear.

To investigate this, 30 patients with rotator cuff tendinopathy and 30 healthy subjects will be evaluated before and immediately after performing the exercise. Three measurements will be done: ultrasonographic measurement of tendon thickness, power Doppler imaging and measurement of microcirculation around the tendon with Oxygen to see. All measurements are non-invasive, pain free and without risks for the human body.

ELIGIBILITY:
Inclusion Criteria Patients:

* Male/ Female
* 18-40 years old
* Unilateral shoulder pain for at least 3 months
* Pain of at least 3/10 on a visual analogue scale
* Painful arc or pain at end range abduction
* 2/3 impingement tests positive
* 2/4 resistance tests positive
* Pain at insertion rotator cuff

Exclusion Criteria Patients:

* Spurling test positive
* Shoulder surgery in the past
* Osteoarthritis shoulder
* Full thickness ruptures

Inclusion Criteria Healthy subjects:

* Male/ Female
* 18-40 years old

Exclusion Criteria Healthy subjects:

* Shoulder pain during the last 3 months
* Shoulder surgery in the past
* Neck pain or disability
* Systemic disease (e.g. Marfan, Ehlers Danlos,…)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Tendon thickness measurement | After 30 minutes rest, before performing the exercise.
  Grey scale ultrasound examination is used.
Tendon vascularisation examination. | After 30 minutes rest, before performing the exercise.
  Power Doppler ultrasound examination is used.
Microcirculation around the tendon examination. | After 30 minutes rest, before performing the exercise.
  Oxygen to see (spectrophotometry and laser Doppler) will be used.

SECONDARY OUTCOMES:
Tendon thickness measurements. | 10 minutes after performing the exercise.
  Grey scale ultrasound examination is used.
Tendon vascularisation examination. | 10 minutes after performing the exercise.
  Power Doppler ultrasound examination is used.
Microcirculation around the tendon examination. | 10 minutes after performing the exercise.
  Oxygen to see (spectrophotometry and laser Doppler) will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Ann Cools, MD, PhD, Principal Investigator — University Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium